CLINICAL TRIAL: NCT06056297
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Mavorixafor in Participants With Congenital and Acquired Primary Autoimmune and Idiopathic Chronic Neutropenic Disorders Who Are Experiencing Recurrent and/or Serious Infections
Brief Title: A Study of Mavorixafor in Participants With Congenital and Acquired Primary Autoimmune and Idiopathic Chronic Neutropenic Disorders Who Are Experiencing Recurrent and/or Serious Infections
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X4P-001-110; 2023-508482-32-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Neutropenia
Keywords: Mavorixafor; Chronic neutropenia; Chronic idiopathic neutropenia; Severe Congenital Neutropenia (SCN); C-X-C chemokine receptor 4 (CXCR4); Congenital and acquired neutropenia; Autoimmune disease; Cohen syndrome; Barth syndrome; ELANE; G6PC3; GSD1b; Kostmann disease; Shwachman-Diamond syndrome; Autoimmune neutropenia (AIN)
MeSH Terms: conditions — Neutropenia; Neutropenia, Severe Congenital, Autosomal Recessive 3; Autoimmune Diseases; Cohen syndrome; Barth Syndrome; Shwachman-Diamond Syndrome | interventions — mavorixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavorixafor (Experimental): Participants will receive mavorixafor orally once daily starting from Day 1 through Week 52.
  Interventions: Drug: Mavorixafor
- Placebo (Placebo Comparator): Participants will receive placebo to match mavorixafor orally once daily starting from Day 1 through Week 52.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavorixafor — Mavorixafor will be administered per schedule specified in the arm description.
  Other Names: X4P-001
  Arms: Mavorixafor
Drug: Placebo — Placebo will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and evaluate the safety and tolerability of mavorixafor in participants with congenital or acquired primary autoimmune and idiopathic chronic neutropenic disorders who are experiencing recurrent and/or serious infections as assessed by demonstrating its clinical benefit and increasing levels of circulating neutrophils.

DETAILED DESCRIPTION:
All participants will continue their pre-study background therapy, defined as the participant's current treatment regimen. Options include, but are not limited to, granulocyte-colony stimulating factor (G-CSF), immunoglobulin replacement therapy, prophylactic antibiotics, or "watchful waiting".

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of congenital or acquired primary autoimmune and idiopathic chronic neutropenic disorder ≥6 months prior to the screening visit that is not attributable to medications, active or recent infections or malignancy.
* Congenital Neutropenia, including but not limited to these classifications:

  1. Isolated with a permanent (non-cyclic) presentation, for example, elastase, neutrophil expressed (ELANE), colony stimulating factor 3 receptor (CSF3R), C-X-C chemokine receptor 2 (CXCR2), Wiskott-Aldrich syndrome (WAS)
  2. Associated with extra-hematologic manifestations, for example, Barth syndrome, Cohen syndrome, glucose-6-phosphatase catalytic subunit 3 (G6PC3), Kostmann disease
  3. Associated with metabolic disorders, for example, glycogen storage disease 1b (GSD1b)
  4. Shwachman-Diamond syndrome
* Acquired Primary Neutropenia

  1. Chronic idiopathic neutropenia
  2. Primary autoimmune neutropenia. Other chronic neutropenia (CN) disorders that may be eligible for enrollment can be clarified and approved upon discussion with study Medical Monitor.
* Have an ANC <1000 cells/µL during screening (single ANC value from hematology) and confirmed trough mean ANC (mean value of multiple ANC measurements over 6 hours) at baseline visit, with no clinical evidence of systemic infection.
* Prior history of recurrent and/or serious infections during the 12 months preceding the screening visit (that is, suffering sequelae of chronic neutropenia), as defined by having at least 2 infections in the last 12 months that meet the following criteria:
* Infection requiring the use of antibiotics (intravenous [IV]/oral); OR
* Infection requiring a visit to healthcare facility (including but not limited to emergency room visit, urgent care facility, primary care physician's office, or in-patient hospitalization);

AND for all potential participants:

* Infections considered by the Investigator to be likely related to the potential participant's CN disorder.
* Participants who are on G-CSF or other active background therapy must have been receiving these therapies during the previous 12 months while continuing to suffer from infections, be on a stable dose and dosing schedule for ≥4 weeks prior to screening visit and remain on this dose and dosing schedule throughout the study (unless ANC >10,000 cells/µL for ≥4 weeks).
* Participants must be willing to keep their G-CSF or other background therapy doses/regimens stable (other than for safety reasons) for the duration of the study.

Key Exclusion Criteria:

* A diagnosis of secondary neutropenia including those due to:

  1. Hypersplenism
  2. Infection
  3. Malignancy
  4. Autoimmune disease, for example, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, graft-versus-host disease, thyroid disease
  5. Nutritional deficiency, for example, vitamin B12, folic acid, copper, caloric malnutrition
  6. Drug-induced cause, for example, chemotherapy, clozapine, antiretrovirals, antibiotics, monoclonal antibodies.
* A diagnosis of any of the following:

  1. Aplastic anemia
  2. Warts, hypogammaglobulinemia, infections, and myelokathexis (WHIM) syndrome
  3. Certain CNs, including but not limited to these classifications are excluded:

     1. Isolated with a cyclic presentation, for example, elastase, neutrophil expressed (ELANE)
     2. Associated with immune dysregulation, for example, common variable immunodeficiency (CVID), autoimmune lymphoproliferative syndrome (ALPS), familial hemophagocytic lymphohistiocytosis, Chédiak-Higashi syndrome, GATA-binding protein 2 (GATA2) deficiency syndrome
     3. Associated with bone marrow failure, for example, Fanconi anemia, Diamond-Blackfan anemia
  4. Neutropenia associated with a Duffy-null phenotype (formerly known as benign ethnic neutropenia). However, a participant with an autosomal dominant pathogenic variant in a gene associated with CN on a Duffy-null background may be eligible for inclusion
* A medical or personal condition that may potentially compromise the safety of the participant, may preclude the participant's successful completion of the clinical study, or could, in the opinion of the Investigator or the Medical Monitor, interfere with the objectives of the study.
* Received more than 1 dose of mavorixafor in the past.
* Received C-X-C chemokine receptor 4 (CXCR4) antagonist (other than mavorixafor) in the past 6 months.
* Participants taking pegylated-G-CSF unless they have a diagnosis of congenital neutropenia confirmed at screening.
* Participant is currently taking or has taken other investigational drug <30 days prior to the screening visit or 5 half-lives, whichever is longer.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Co-primary Endpoint: Annualized Infection Rate Based on Infections Adjudicated by Blinded Infection Adjudication Committee (BIAC) During the Treatment Period | Up to 52 Weeks
Co-primary Endpoint: Number of Participants Meeting the Definition of a Positive Absolute Neutrophil Count (ANC) Response | Up to 52 weeks
  Positive ANC response: Increase of ANC >500 cells/microliter (µL) from baseline.

SECONDARY OUTCOMES:
Infection Severity Based on Common Terminology Criteria for Adverse Events (CTCAE) Adjudicated by a BIAC During the Treatment Period | Up to 52 Weeks
Infection Duration Based on Duration of Infections Adjudicated by a BIAC During the Treatment Period in Those Participants who Developed Infections | Up to 52 Weeks
Antibiotic Use Due to Infection, Characterized by the Frequency of Antibiotic Use During the Treatment Period | Up to 52 Weeks
Oral Ulcers, as Assessed by Presence or Absence of Ulcers During the Treatment Period | Up to 52 Weeks
Change From Baseline in Patient Reported Outcomes Measurement Information System Short Form (PROMIS SF) Fatigue Questionnaire Total Score | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Global Head of Clinical Development and Safety, Study Director — X4 Pharmaceuticals
Locations (104):
- United States (19):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UC Irvine, Irvine, California
  - Orso Health, La Jolla, California
  - University of California, Los Angeles-UCLA, Los Angeles, California
  - Orso Health, Torrance, California
  - University of Southern Florida, St. Petersburg, Florida
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital/ Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Froedtert And Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital El Cruce, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Santorio 9 de Julio, San Miguel de Tucumán
- Australia (3):
  - Perth Children's Hospital, Nedlands
  - Icon Cancer Centre Southport, Southport
  - Ballarat Oncology And Haematology Services, Wendouree
- University of Alberta Hospital, Edmonton, Canada
- Clinica IMBANACO S.A.S, Cali, Colombia
- Czechia (2):
  - The University Hospital Brno, Brno
  - Motol University Hospital, Prague
- France (6):
  - Institute of Hematology and Pediatric Oncology - Lyon, Lyon
  - Hôpital Saint Louis, Paris
  - Hospital Armand Trousseau Ap-Hp, Paris
  - Hôpital Necker - Enfants Malade, Paris
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Institut Universitaire de Cancérologie de Toulouse - Oncopôle, Toulouse
- Georgia (4):
  - LTD "Israeli-Georgian Medical Research Clinic Healthycore", Tbilisi
  - LEPL The First University Clinic of Tbilisi State Medical University, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - LTD Multiprofile Clinic Concilium Medulla, Tbilisi
- Germany (2):
  - Klinik und Poliklinik fur Kinder- und Jugendmedizin, Universitatsklinikum Carl Gustav Carus an der TU, Dresden
  - Universitaetsklinikum Carl Gustav Carus Tu Dresden, Dresden
- Greece (4):
  - Hellenic Airforce 251 General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - The Olympion Private General Clinic, Pátrai
  - AHEPA General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - CMC Deli Klinika, Budapest
  - Semmelweis University, Budapest
  - Teaching Hospital Markusovszky, Szombathely
- India (4):
  - Indira Gandhi Institute Of Medical Sciences, Patna, Bihar
  - Nirmal Hospital Private Limited, Surat, Gujarat
  - Pacific Medical College and Hospital, Udaipur, Rajasthan
  - Yashoda Hospital, Hyderabad, Telangana
- Israel (4):
  - Ruth Rappaport Children's Hospital, Rambam Health Corporation, Haifa
  - Hadassah University Hospital-ein Kerem, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (6):
  - A. O. U. delle Marche, Torrette, Ancona
  - ASST Spedali Civili di Brescia, Brescia
  - IRCCS Instituto G. Gaslini, Genova
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori (IRST) Dino Amadori, Meldola
  - IRCCS San Gerardo Dei Tintori, Monza
  - Bambino Gesu Children's Hospital, Roma
- Hospital Pakar Kanak-Kanak UKM, Kuala Lumpur, Malaysia
- Portugal (4):
  - Unidade Local de Saúde da Região de Aveiro, Aveiro
  - Unidade Local de Saude Coimbra - Paediatric Hospital, Coimbra
  - Unidade Local de Saude Coimbra - Quinta dos Vales, Coimbra
  - Unidade Local de Saude Santa Maria, Lisbon
- Romania (4):
  - Spitalul Clinic Colentina Site 1, Bucharest
  - Spitalul Clinic Colentina Site 2, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Județean de Urgență, Târgu Mureş
- University Clinical Centre of Serbia, Belgrade, Serbia
- Spain (11):
  - ICO Badalona - Institut Català d'Oncologia, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital San Pedro De Alcantara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital De La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico de la Fe, Valencia
- Switzerland (2):
  - Inselspital - University Hospital Bern Site 1, Bern
  - Inselspital - University Hospital Bern Site 2, Bern
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (5):
  - Namik Kemal University (Tekirdağ Namık Kemal Üniversitesi), Tekirdağ, Süleymanpaşa
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training And Research Hospital, Ankara
  - Ankara University School of Medicine, Ankara
  - Uludag University Faculty Of Medicine, Nilufer
  - Ondokuz Mayis University Medical Faculty Hospital, Samsun
- Ukraine (6):
  - Lviv Regional Clinical Diagnostic Centre, Lviv, Oblast
  - Medical Center Dobrobut-Clinic LLC, Kyiv
  - Medical Center Ok Clinic of International Institute of Clinical Research LLC, Kyiv
  - Llc Onto-Med, Kyiv
  - Communal non-commercial enterprise "Ternopil City Children's Communal Hospital", Ternopil
  - Medical Center The Clinic of Hospodarskyy LLC, Ternopil
- United Kingdom (6):
  - University Hospital of Wales, Cardiff
  - Cardiff And Vale University Health Board, London
  - Royal Free London Nhs Foundation Trust Royal Free Hospital, London
  - King's College Hospital, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - Great Ormond street Hospital for Children NHS Trust, London

IPD SHARING:
Plan to Share IPD: No